CLINICAL TRIAL: NCT06852989
Title: Shared Interactive Book Reading in Preschool Children With Neurodevelopmental Disorders: Effects on Language Development and Reading Habits
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: SIBR-PN
Record Dates: First submitted 2025-02-19; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Neurodevelopmental Disorders; Autism Spectrum Disorder; Intellectual Disabilities; Language Disorders in Children
Keywords: shared reading; early literacy; neurodevelopmental disorder; autism; intellectual disability; vocabulary; shared reading habits; language disorders; shared interactive book reading
MeSH Terms: conditions — Neurodevelopmental Disorders; Autism Spectrum Disorder; Intellectual Disability; Literacy; Autistic Disorder; Language Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study group: 27 children with neurodevelopmental disorders
  Interventions: Other: Shared book reading intervention
- Comparison group: 26 children with neurodevelopmental disorders

INTERVENTIONS:
Other: Shared book reading intervention — The study group participated in a parent training program focusing on shared interactive reading practices and attended nine read-aloud meetings with their children under the supervision of a trained librarian.
  Other Names: Parent-based book reading intervention
  Groups: Study group

SUMMARY:
The goal of this observational retrospective study is to explore the effects of a parent-based book reading intervention on children with neurodevelopmental disorders. The project consisted of interactive lessons for parents and shared reading experiences. It took place between May 2021 and June 2022 in Rome and at the time children were receiving neuropsychomotor and speech therapy sessions based on the developmental profile.

The investigators'primary goal is to investigate lexical quotients of children who participated in the project to explore whether it had an impact on their language development. The secondary goal is to assess shared reading habits.

For both outcome measures, researchers will compare the group who partecipated in the study with a cohort of children with the same characteristics who also attended Fondazione Don Carlo Gnocchi for rehabilitation purposes.

Patients and their family will not be asked for any further engagement because all data will be taken from medical records.

ELIGIBILITY:
Inclusion criteria for the study group:

* age between 1 and 6 years old
* having attended at least 2 out of 5 parent training meetings and 2 out of 9 reading aloud sessions
* at least one caregiver with a good command of the Italian language,
* having given written consent to participate

Exclusion Criteria for both groups:

* cerebral palsy or severe sensory disorder (deafness, blindness)
* limited command of the italian language
* lack of informed consent

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preschool children with neurodevelopmental disorders attending Fondazione Don Carlo Gnocchi's rehabilitation center
Sampling Method: Non-Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Lexical quotients (receptive and expressive) | February 2025 - August 2025
  We will analyze receptive and expressive lexical quotient of both study and comparison group.

SECONDARY OUTCOMES:
Non-standardized shared-reading habits questionnaire | February 2025 - August 2025
  We will analyze the impact of the project on families' shared reading habits through a custom-built self-administered questionnaire. The questionnaire has been delivered at the beginning and at the end of the project.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Iuvone, Doctor, Principal Investigator — Fondazione Don Carlo Gnocchi Onlus
Locations (1):
- Fondazione Don Carlo Gnocchi Onlus, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided